CLINICAL TRIAL: NCT02978794
Title: Implementation of Clinical Pathway to Improve Quality of Healthcare in Stroke Inpatients
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Changhua Christian Hospital (Other)
Responsible Party: Principal Investigator, Ta-Sen Wei,MD, Director, Physical Medical and Rehabilitation, Principal Investigator,, Changhua Christian Hospital
Other Study IDs: CCH-161006
Record Dates: First submitted 2016-11-29; First posted 2016-12-01 (Estimated); Last update posted 2021-07-01 (Actual); Status verified 2021-06

CONDITIONS: Stroke
Keywords: stroke, clinical pathway, medical care
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
With the extension of the average life expectancy, the incidence of cardiovascular diseases is also rising. Stroke in Taiwan has been the leading cause of morbidity and mortality, but also in countries around the world), stroke and the impact of socio-economic and health spending are large how to reduce the degree of disability after stroke is an important issue in medicine. For a long time, the resident will fill the clinical pathway form before the stroke inpatients were discharged. We also analyzed the data of clinical pathway every three months.

According to the current data of stroke clinical pathway included demographic data, length of hospitalization days, complications, functional independent measure, Brunnstrom motor recovery stage, mini-mental state examination, geriatric depression scale, blood pressure data, and post-stroke checklist for a retrospective analysis to provide more complete and more comprehensive information on follow-up care for stroke patients and effective use of medical resources, to improve the quality of future medical care and quality of life for stroke patients.

ELIGIBILITY:
Inclusion Criteria:

1. Ischemic and hemorrhagic stroke patients
2. MRI confirmed the diagnosis of stroke
3. Within three months of onset of unilateral limb hemiplegia in patients

Exclusion Criteria:

1. Initial tracheostomy impantation and hospital stay is less than 5 days
2. Combined with other neurological diseases, such as epilepsy, multiple neuropathy, Meniere's disease, vestibular neuritis, Parkinson's disease, dementia or cerebellar atrophy, etc.
3. Significant lesions of the lower limb joints, including joint contractures, lower limb fractures, joint replacement or long-term pain in patients with osteoarthritis
4. Unstable signs of life (if not through the tilt bed test) or severe cardiopulmonary disease
5. Those who can not cooperate with the study or who have not signed the inform consent

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: stroke inpatient
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2016-11; Primary Completion 2022-02 (Estimated); Study Completion 2022-02 (Estimated)

PRIMARY OUTCOMES:
functional independent measurement | 1 year
post-stroke checklist | 1 year
Brunnstrom motor recovery stage | 1 year